CLINICAL TRIAL: NCT00747123
Title: A Phase 2a, Multi-Center, Randomized, Multiple-Dose Study to Evaluate the Safety, Tolerability and Efficacy of ACE-011 (hActRIIA-IgG1) in Patients With Osteolytic Lesions of Multiple Myeloma
Brief Title: A Safety, Tolerability and Efficacy Study of ACE-011 in Patients With Osteolytic Lesions of Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A011-04
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ACE-011

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Subcutaneous injection on days 1, 29, 57 and 85.
  Interventions: Biological: Placebo
- ACE-011 0.1 mg/kg (Experimental): Subcutaneous injection of ACE-011 0.1 mg/kg every 28 days totaling four doses (days 1, 29, 57 and 85).
  Interventions: Biological: ACE-011
- ACE-011 0.3 mg/kg (Experimental): Subcutaneous injection of ACE-011 0.3 mg/kg every 28 days totaling four doses (days 1, 29, 57 and 85).
  Interventions: Biological: ACE-011
- ACE-011 0.5 mg/kg (Experimental): Subcutaneous injection of ACE-011 0.5 mg/kg every 28 days totaling four doses (days 1, 29, 57 and 85).
  Interventions: Biological: ACE-011

INTERVENTIONS:
Biological: ACE-011 — ACE-011 given by the subcutaneous route of administration monthly for 4 doses.
  Other Names: hActRIIA-IgG1
  Arms: ACE-011 0.1 mg/kg; ACE-011 0.3 mg/kg; ACE-011 0.5 mg/kg
Biological: Placebo — Placebo given by the subcutaneous route of administration monthly for 4 doses.
  Arms: Placebo

SUMMARY:
Multi-center, randomized, multiple-dose study to evaluate the safety, tolerability and efficacy of ACE-011 in patients with osteolytic lesions of multiple myeloma.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient at least 18 years of age with stage II or III multiple myeloma
* One or more lytic bone lesions
* If currently receiving bisphosphonate therapy, have been on a stable dose for ≥ 2 months before dosing day 1 or must not have received bisphosphonates within 2 months of dosing day 1
* If patient has undergone previous autologous or allogenic hematopoietic stem cell transplantation (HSCT), they must be stable (in the opinion of the investigator) and be a minimum of 6 months since HSCT
* Has planned HSCT for the duration of the study
* Has moles or lesions that are currently undiagnosed, but are suspect for malignancy
* Has an underlying condition that may result in abnormal bone metabolism other than cancer related bone lesions, such as a history of hyperparathyroidism, hypoparathyroidism, hypocalcemia, rheumatoid arthritis, myeloproliferative disorder, gout, Paget's disease of the bone, or osteomalacia; patients with a diagnosis of osteoporosis prior to multiple myeloma diagnosis are eligible to participate.

Key Exclusion Criteria:

* Known underlying condition that may result in abnormal bone metabolism other than cancer related bone lesions
* History of polyneuropathy ≥ grade 3
* Patients with plasma cell leukemia
* Planned stem cell transplant (HSCT) or radiation for the duration of the study
* Skeletal related event within 2 weeks of study enrollment
* Has received erythropoiesis-stimulating agents (ESAs) within the last 21 days or is planned to receive ESAs during the course of the study
* Has received anti-myeloma therapy within the last 21 days
* Is scheduled to receive local radiation to bone during the course of the study
* Has taken estrogen, androgen, anabolic steroids, calcitonin or other bone-active drugs within 4 months of study enrollment
* Woman of childbearing potential (not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2009-08-01 (Actual); Study Completion 2009-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abderrahmane Laadem, MD, Study Director — Celgene Corporation
Locations (2):
- Russia (2):
  - Investigative Site, Moscow
  - Investigative Site, Saint Petersburg

REFERENCES:
- [Background] Abdulkadyrov KM, Salogub GN, Khuazheva NK, Sherman ML, Laadem A, Barger R, Knight R, Srinivasan S, Terpos E. Sotatercept in patients with osteolytic lesions of multiple myeloma. Br J Haematol. 2014 Jun;165(6):814-23. doi: 10.1111/bjh.12835. Epub 2014 Mar 21. PMID 24650009

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo was administered within 28 days of screening. Subsequent doses were administered every 28 days for a total of four doses.
- 0.1 mg/kg ACE 011: 0.1 mg/kg administered via subcutaneous injection every 28 days for a total of four doses (i.e., Days 1, 29, 57, and 85), with safety follow-up visits 1 week after each dose (i.e., Days 8, 36, 64, and 92). After completion of the treatment period, participants returned to the study site monthly for follow-up assessments for an additional 3 months (i.e., Days 113, 141, and 169).
- 0.3 mg/kg ACE 011: 0.3 mg/kg administered via subcutaneous injection every 28 days for a total of four doses (i.e., Days 1, 29, 57, and 85), with safety follow-up visits 1 week after each dose (i.e., Days 8, 36, 64, and 92). After completion of the treatment period, participants returned to the study site monthly for follow-up assessments for an additional 3 months (i.e., Days 113, 141, and 169)
- 0.5 mg/kg ACE 011: 0.5 mg/kg administered via subcutaneous injection every 28 days for a total of four doses (i.e., Days 1, 29, 57, and 85), with safety follow-up visits 1 week after each dose (i.e., Days 8, 36, 64, and 92). After completion of the treatment period, participants returned to the study site monthly for follow-up assessments for an additional 3 months (i.e., Days 113, 141, and 169).
Period: Overall Study
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011
Started | 6 | 8 | 8 | 8
Completed | 6 | 6 | 7 | 7
Not Completed | 0 | 2 | 1 | 1
Not completed — Investigator's request | 0 | 0 | 1 | 0
Not completed — Withdrew consent | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011 | Total
Number analyzed (Participants) | 6 | 8 | 8 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (7.92) | 60.5 (13.28) | 63.6 (7.50) | 57.8 (12.30) | 60.9 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 4 | 15
  Male | 2 | 6 | 3 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 7 | 8 | 8 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A treatment emergent adverse event (TEAE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causality assessment. A TEAE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. Any worsening (i.e., any clinical significant adverse change in frequency and/or intensity) of a preexisting condition, which was temporally associated with the use of the sponsor's medicinal (investigational) product, was also a TEAE. The number of participants with at least one TEAE are reported.
Time Frame: From first dose to termination visit on Day 169
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011
Number analyzed (Participants) | 6 | 8 | 8 | 8
Participants | 4 | 7 | 7 | 8

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Related to Study Drug
Description: A treatment emergent adverse event (TEAE) related to study drug was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, that was determined to be related to the study drug. A TEAE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. Any worsening (i.e., any clinical significant adverse change in frequency and/or intensity) of a preexisting condition, which was temporally associated with the use of the sponsor's medicinal (investigational) product, was also a TEAE. The number of participants with at least one TEAE are reported. Treatment emergent adverse events were assessed by the investigator as possibly, probably, or definitely related to the study drug.
Time Frame: From first dose to termination visit on Day 169
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011
Number analyzed (Participants) | 6 | 8 | 8 | 8
Participants | 0 | 1 | 0 | 1

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) was defined as any untoward medical occurrence that at any dose (including overdose) that was fatal, was life threatening, required or prolonged inpatient hospitalization, resulted in permanent or significant disability/incapacity, or was a congenital anomaly/birth defect. The number of participants with at least one serious adverse event are reported.
Time Frame: From first dose up to termination visit on Day 169
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011
Number analyzed (Participants) | 6 | 8 | 8 | 8
Participants | 0 | 1 | 0 | 3

4. Primary Outcome: Change From Baseline in Hemoglobin
Description: Summary of the change from baseline in hemoglobin (g/dL) by the pre-specified timepoints. Baseline was defined as the last measurement prior to dosing. Data were summarized for all treated participants who had at least 1 postdosing measurement.
Time Frame: Day 1 (baseline), Day 8, Day 29, Day 36, Day 57, Day 85, Day 113, Day 169
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011
Number analyzed (Participants) | 6 | 8 | 8 | 8
g/dL
  Day 8 | 0.47 (0.288) | 0.89 (1.254) | 0.83 (0.599) | 0.80 (0.844)
  Day 29: number analyzed (Participants) | 6 | 7 | 8 | 7
  Day 29 | 0.50 (0.607) | -0.91 (1.844) | 0.66 (0.457) | 0.96 (1.648)
  Day 36: number analyzed (Participants) | 6 | 8 | 8 | 6
  Day 36 | 1.02 (0.643) | 0.73 (1.873) | 1.00 (0.787) | 1.48 (1.167)
  Day 57: number analyzed (Participants) | 6 | 7 | 8 | 7
  Day 57 | 0.53 (0.602) | 0.47 (1.682) | 1.09 (1.022) | 1.00 (1.22)
  Day 85: number analyzed (Participants) | 6 | 7 | 8 | 7
  Day 85 | 0.78 (0.958) | 0.57 (0.907) | 0.86 (1.323) | 1.56 (0.704)
  Day 113: number analyzed (Participants) | 6 | 6 | 8 | 7
  Day 113 | 0.33 (0.789) | 0.53 (1.141) | 0.96 (1.620) | 0.97 (1.024)
  Day 169/Early Termination: number analyzed (Participants) | 6 | 6 | 8 | 7
  Day 169/Early Termination | 0.13 (1.140) | 0.57 (1.500) | 0.33 (1.763) | 0.03 (2.392)

5. Primary Outcome: Number of Participants With Electrocardiogram Abnormalities
Description: The number of participants with at least one clinically significant postbaseline electrocardiogram abnormality. The abnormalities included left ventricular hypertrophy, atrial fibrillation, sinus bradycardia, sinus tachycardia, and myocardial ischemia. Data is reported as the cumulative number of participants with abnormalities over the scheduled collection timepoints.
Time Frame: Pre-dose, Day 1, Day 92, and Day 169
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011
Number analyzed (Participants) | 6 | 8 | 8 | 8
Participants | 4 | 2 | 2 | 2

6. Primary Outcome: Number of Participants With Hypertension or Increased Blood Pressure
Description: The number of participants who experienced hypertension or an increase in blood pressure from baseline up to Day 92. Abnormal blood pressure was defined as:
  * Systolic blood pressure ≤ 90 or ≥ 180 mmHg
  * Systolic blood pressure change (increase or decrease) ≥ 20 mmHg
  * Diastolic blood pressure ≤ 60 or ≥ 100 mmHg
  * Diastolic blood pressure change (increase or decrease) ≥ 15 mmHg
Time Frame: From baseline up to Day 92
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011
Number analyzed (Participants) | 6 | 8 | 8 | 8
Participants | 0 | 1 | 0 | 2

7. Secondary Outcome: Number of Participants With Skeletal-related Events (SRE)
Description: Skeletal-related events are defined as pathologic fracture, radiation therapy to bone, surgery to bone, or spinal cord compression, within 2 weeks of study enrollment. They are determined by skeletal surveys, including x-rays of the skull, entire spine, pelvis, ribs, humeri, and femora.
Time Frame: From first dose up to 2 weeks post first dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011
Number analyzed (Participants) | 6 | 8 | 8 | 8
Participants | 0 | 1 | 2 | 2

8. Secondary Outcome: Percent Change From Baseline in Bone Pain Visual Analog Scale (VAS)
Description: The visual analog scale (VAS) is a pain rating scale. Scores are based on the percent change from baseline (Day 1) in self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm). Measurements from the starting point (left end) of the scale to the patients' marks are recorded in centimeters and are interpreted as their pain. The values can be used to track pain progression for a patient or to compare pain between patients with similar conditions. In addition to pain, the scale has also been used to evaluate mood, appetite, asthma, dyspepsia, and ambulation.
Time Frame: From baseline (Day 1) to Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: All treated participants who had at least 1 postdosing measurement
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | 0.1 mg/kg ACE 011 | 0.3 mg/kg ACE 011 | 0.5 mg/kg ACE 011
Number analyzed (Participants) | 6 | 8 | 8 | 7
Percent change
  Day 29 | -6.0 (12.25) | -9.4 (22.60) | -5.8 (25.03) | -6.4 (23.87)
  Day 57: number analyzed (Participants) | 6 | 7 | 8 | 7
  Day 57 | -7.2 (6.77) | -8.0 (26.09) | -11.0 (33.87) | -11.6 (26.34)
  Day 85: number analyzed (Participants) | 6 | 7 | 8 | 7
  Day 85 | -4.5 (3.78) | -12.7 (23.08) | -10.5 (37.50) | -11.1 (28.79)
  Day 113: number analyzed (Participants) | 6 | 6 | 8 | 7
  Day 113 | -3.5 (4.46) | -13.7 (25.03) | -12.3 (38.04) | -11.4 (29.43)
  Day 141: number analyzed (Participants) | 6 | 6 | 8 | 7
  Day 141 | 0.7 (13.05) | -13.7 (25.26) | -15.0 (37.33) | -12.1 (32.79)
  Day 169: number analyzed (Participants) | 6 | 6 | 8 | 7
  Day 169 | -3.0 (7.59) | -14.7 (24.59) | -15.0 (38.40) | -13.6 (30.36)

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 10 months). SAEs and Other AEs were assessed from first dose to Day 169.
Groups:
- ACE 011 0.1 mg/kg: 0.1 mg/kg administered via subcutaneous injection every 28 days for a total of four doses (i.e., Days 1, 29, 57, and 85), with safety follow-up visits 1 week after each dose (i.e., Days 8, 36, 64, and 92). After completion of the treatment period, participants returned to the study site monthly for follow-up assessments for an additional 3 months (i.e., Days 113, 141, and 169).
- ACE 011 0.3 mg/kg: 0.3 mg/kg administered via subcutaneous injection every 28 days for a total of four doses (i.e., Days 1, 29, 57, and 85), with safety follow-up visits 1 week after each dose (i.e., Days 8, 36, 64, and 92). After completion of the treatment period, participants returned to the study site monthly for follow-up assessments for an additional 3 months (i.e., Days 113, 141, and 169)
- ACE 011 0.5 mg/kg: 0.5 mg/kg administered via subcutaneous injection every 28 days for a total of four doses (i.e., Days 1, 29, 57, and 85), with safety follow-up visits 1 week after each dose (i.e., Days 8, 36, 64, and 92). After completion of the treatment period, participants returned to the study site monthly for follow-up assessments for an additional 3 months (i.e., Days 113, 141, and 169).
Arm/Group | ACE 011 0.1 mg/kg | ACE 011 0.3 mg/kg | ACE 011 0.5 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/8 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 3/8 | 0/6
Other Adverse Events (participants affected / at risk) | 7/8 | 7/8 | 8/8 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACE 011 0.1 mg/kg (N=8) | ACE 011 0.3 mg/kg (N=8) | ACE 011 0.5 mg/kg (N=8) | Placebo (N=6)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACE 011 0.1 mg/kg (N=8) | ACE 011 0.3 mg/kg (N=8) | ACE 011 0.5 mg/kg (N=8) | Placebo (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 6 | 6 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial conduction time prolongation (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.